CLINICAL TRIAL: NCT03136055
Title: A Pilot Study of Pembrolizumab-based Therapy in Previously Treated High Grade Neuroendocrine Carcinomas
Brief Title: Pembrolizumab-based Therapy in Previously Treated High Grade Neuroendocrine Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 169524; NCI-2017-01728 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-04-18; First posted 2017-05-02 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: High Grade Malignant Neuroendocrine Carcinoma (Diagnosis)
Keywords: NEC
MeSH Terms: conditions — Disease | interventions — pembrolizumab; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: Pembrolizumab only (Experimental): Participants will receive 200 mg of pembrolizumab via IV over 30 minutes every 3 weeks for 24 months or 35 administrations (whichever comes first).
  Interventions: Drug: Pembrolizumab
- Part B: Pembrolizumab + Chemotherapy (Experimental): Participants will receive 200 mg of pembrolizumab via IV over 30 minutes every 3 weeks for 24 months or 35 administrations (whichever comes first) and chemotherapy treatment of 125 mg/m^2 of irinotecan via IV on days 1 and 8 of each 21-day cycle or paclitaxel via IV on days 1, 8, and 15 of each 21-day cycle per physician discretion
  Interventions: Drug: Pembrolizumab; Drug: Irinotecan; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Given Intravenously (IV)
  Other Names: Keytruda
Drug: Irinotecan — Given IV
  Other Names: Camptosar
  Arms: Part B: Pembrolizumab + Chemotherapy
Drug: Paclitaxel — Given IV
  Other Names: Taxol
  Arms: Part B: Pembrolizumab + Chemotherapy

SUMMARY:
This is a pilot study of pembrolizumab-based therapy in previously treated extrapulmonary poorly differentiated neuroendocrine carcinoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. Evaluate the best overall response rate (ORR) of pembrolizumab or pembrolizumab plus chemotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (investigator-reported).

SECONDARY OBJECTIVE:

1. To determine the safety and tolerability of pembrolizumab-based therapy in this patient population.
2. To evaluate duration of response (DOR) in participants receiving pembrolizumab or pembrolizumab plus chemotherapy.
3. To evaluate progression free survival (PFS) in participants treated with pembrolizumab or pembrolizumab plus chemotherapy (median PFS and 18 wk PFS).
4. To evaluate overall survival (OS) in participants receiving pembrolizumab or pembrolizumab plus chemotherapy.

OUTLINE:

Part A: Participants are treated with pembrolizumab alone. An adaptive Simon's two-stage design was used, and the overall plan hinges on the activity of single agent pembrolizumab in the first stage of Part A. If there is sufficient activity in the first stage of Part A, the study will expand to the second stage of Part A and forgo Part B. If there is insufficient activity in the first stage of Part A, the study will proceed to the first stage of Part B (pembrolizumab plus chemotherapy).

Part B: Participants are treated with pembrolizumab plus chemotherapy (physician's choice, paclitaxel or irinotecan). Patients with stable disease (SD) or better after 9 cycles (27 weeks) of pembrolizumab-based therapy will have the option to continue with pembrolizumab alone, unless the first partial response (PR) or complete response (CR) is noted at 27 weeks.

All participants will undergo a pre-treatment tumor biopsy (unless the tumor is inaccessible and/or a biopsy is not felt to be in the participant's best interest). Participants may continue study treatment until progressive disease (PD), unacceptable adverse events, inter-current illness that prevents further administration of treatment, investigator's decision to withdraw the participant, the participant withdraws consent, pregnancy of the participant, noncompliance with trial treatment or procedure requirements, participant receives 35 treatments (approximately 2 years) of pembrolizumab, or administrative reasons requiring cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. Have a histologically proven locally advanced or metastatic high grade (G3) poorly differentiated neuroendocrine carcinoma (NEC).

   1. Includes small cell and large cell neuroendocrine carcinoma of unknown primary or any extrapulmonary site (and poorly differentiated NEC, not otherwise specified)
   2. Includes neuroendocrine prostate cancer (de novo or treatment-emergent) of prostate if small cell or large cell histology (histologic evidence of both adenocarcinoma and neuroendocrine carcinoma may be present in same patient).
   3. Other mixed tumors, e.g. mixed neuroendocrine neoplasms (MINENs) with NEC plus adenocarcinoma, squamous or acinar cell component are allowed if the high grade (small or large cell) NEC component comprises >50% of the original sample or subsequent biopsy.
4. Have progressed during or after completion of first line systemic chemotherapy.

   1. No limit to the number of prior chemotherapy regimens.
   2. Early progression on/after adjuvant chemotherapy counts as firstline therapy.
5. Have at least one measurable disease based on RECIST 1.1.
6. Patients must agree to have a biopsy of primary tumor or metastatic tissue at baseline, and there must be a lesion that can be biopsied with acceptable clinical risk (as judged by the investigator).

   1. Patients with unsuccessful baseline biopsies may undergo an additional biopsy attempt (at the same or a different site, determined by the investigator).
   2. For patients with an intact primary and no metastatic site that can be safely biopsied, biopsy of the primary is acceptable, but must be approved by the principal investigator.
   3. Baseline tumor biopsy may be omitted if the tumor is inaccessible and/or a biopsy is not thought to post exceptionally high procedural risk due to location or other factors
7. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Have a life expectancy of greater than 3 months.
9. Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation.

   * Absolute neutrophil count (ANC) >=1,500 /microliter (mcL)
   * Platelets >=100,000 / mcL
   * Hemoglobin >= 9 g/dL or >=5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
   * Serum creatinine OR Measured or calculated creatinine clearance (CrCl) (Creatinine clearance should be calculated per institutional standard. Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl <=1.5 X upper limit of normal (ULN) OR >=60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin <= 1.5 X ULN OR Direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 ULN
   * aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) <=2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin >2.5 g/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) <=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
    * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Has Merkel cell carcinoma, small cell lung carcinoma, or large cell NEC of lung

   * Intermediate grade neuroendocrine tumors are excluded
   * Well differentiated Grade 3 neuroendocrine tumors are excluded
   * Metastatic high-grade prostate carcinoma with evidence of focal neuroendocrine differentiation on prostate biopsy (e.g., positive chromogranin staining by immunohistochemistry) without small cell or large cell NEC morphology are excluded, as are neuroendocrine prostate cancers with phenotype intermediate between adenocarcinoma and small cell
   * Atypical and typical bronchial carcinoids and well differentiated G1 and G2 gastroenteropancreatic (GEP) neuroendocrine tumors (NET) (GEP NETs) are excluded.
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency
4. Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

   - Physiologic doses of steroids (e.g. =< 10 mg prednisone/day or equivalent) are allowed
5. Has a known history of active Bacillus Tuberculosis (TB).
6. History of or high suspicion of Gilbert's disease (safety run-in, Part B only)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
9. Documented progression on and/or intolerance/hypersensitivity to both paclitaxel and irinotecan (Part B only)
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., <= Grade 1 or at baseline) from adverse events due to a previously administered agent.

    * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
    * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
    * Concurrent somatostatin analog therapy is allowed (for control of hormone excess) provided patient has been on stable dose for at least two months and tumor progression has been documented
    * Continuation of androgen deprivation therapy (ADT) allowed for patients with neuroendocrine prostate cancer (in the setting of castration-resistant prostate cancer, CRPC)
11. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with asymptomatic suspected brain metastases (or small lesions of uncertain significance) <1 cm that do not require focal therapy are eligible. (Follow up imaging will be allowed on study, and focal radiation with continuation of protocol therapy allowed if there is progressive disease in the brain and systemic imaging shows stable disease/response).

    - Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks and any neurologic symptoms have returned to baseline), they have no evidence of new or enlarging brain metastases (confirmed by imaging within 28 d of the first dose of trial treatment), and they are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    - Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a history of (non-infectious) pneumonitis/ interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
19. Has received prior therapy with an anti-Programmed Death 1 (PD-1), anti-Programmed Death Ligand 1 (PD-L1), or anti-PD-L2 agent.
20. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
21. Has known active Hepatitis B virus (e.g., HBsAg reactive) or Hepatitis C virus (HCV)(e.g., HCV RNA [qualitative] is detected).
22. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Bergsland, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raj N, Chan JA, Wang SJ, Aggarwal RR, Calabrese S, DeMore A, Fong L, Grabowsky J, Hope TA, Kolli KP, Mulvey CK, Munster PN, Perez K, Punn S, Reidy-Lagunes D, Von Fedak S, Zhang L, Bergsland EK. Pembrolizumab alone and pembrolizumab plus chemotherapy in previously treated, extrapulmonary poorly differentiated neuroendocrine carcinomas. Br J Cancer. 2023 Aug;129(2):291-300. doi: 10.1038/s41416-023-02298-8. Epub 2023 May 19. PMID 37208512

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
Started | 14 | 22
Completed | 14 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy | Total
Number analyzed (Participants) | 14 | 22 | 36
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 2 | 3
  40-49 years old | 2 | 3 | 5
  50-59 years old | 3 | 7 | 10
  60-69 years old | 2 | 5 | 7
  70-79 years old | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 9 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 19 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 22 | 36
Received prior platinum-based therapy [Count of Participants; unit: Participants] — Platinum-based antineoplastic drugs (informally called platins) are chemotherapeutic agents used to treat cancer.
  Participants | 14 | 22 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants in the analysis population who demonstrated complete response (CR) or partial response (PR) radiographically according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by investigator. The analysis will include all subjects treated (ITT) who received at least one dose of the study treatment. If the final study consists of both Part A and Part B, the analysis will be done separately for each part.
Time Frame: Approximately 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 14 | 22
percentage of participants | 7 [0.02 to 33.9] | 5 [0 to 22.8]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first day of study treatment with protocol therapy to the date of death due to any cause. Kaplan-Meier method will be used to summarize OS. Median OS and its 95% confidence interval will be obtained for Part A and B (if available) separately.
Time Frame: Over the duration of the study, which is estimated to be approximately 32 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 14 | 22
months | 7.8 [3.1 to NA] — There were insufficient number of events so the upper limit of the confidence interval could not be calculated. | 4.8 [4.1 to 8.2]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response is defined as the time from the date of first response (CR or PR) until the date of disease progression or death. Duration of response will be reported for Part A and B (if available) separately. Only patients who have a demonstrated response will be used in final analysis.
Time Frame: Over the duration of the study, which is estimated to be approximately 32 months.
Population: Only 1 participant in Part A, and 1 participant in Part B obtained CR or PR
Measure: Number; unit: months
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 1 | 1
months | 18.9 | 6.71

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time from the first day of study treatment with protocol therapy to the date of documented tumor progression or death due to any cause, whichever occurs first, as determined by RECIST v1.1 for PFS. Subjects who did not progress or die will be censored on the date of their last evaluable tumor assessment. Kaplan-Meier method will be used to summarize progression median PFS with 95% confidence interval for Part A and B (if available) separately.
Time Frame: Over the duration of the study, which is estimated to be approximately 32 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 14 | 22
months | 1.8 [1.7 to 21.4] | 2 [1.9 to 3.4]

ADVERSE EVENTS:
Time Frame: Up to 32 months
Arm/Group | Part A: Pembrolizumab Only | Part B: Pembrolizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 11/14 | 21/22
Serious Adverse Events (participants affected / at risk) | 1/14 | 6/22
Other Adverse Events (participants affected / at risk) | 14/14 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pembrolizumab Only (N=14) | Part B: Pembrolizumab + Chemotherapy (N=22)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pembrolizumab Only (N=14) | Part B: Pembrolizumab + Chemotherapy (N=22)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 10 (11)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 12 (20)
Nausea (Gastrointestinal disorders) | 4 (4) | 10 (11)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (9)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (11) | 15 (23)
Pain (General disorders) | 5 (6) | 4 (6)
Fever (General disorders) | 0 (0) | 6 (7)
Edema limbs (General disorders) | 2 (2) | 3 (4)
Infusion related reaction (General disorders) | 2 (3) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (57) | 15 (55)
Neutrophil count decreased (Investigations) | 0 (0) | 9 (11)
Alkaline phosphatase increased (Investigations) | 3 (8) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 4 (10) | 2 (3)
Weight loss (Investigations) | 2 (2) | 4 (5)
Creatinine increased (Investigations) | 3 (10) | 2 (4)
Platelet count decreased (Investigations) | 2 (5) | 3 (4)
White blood cell decreased (Investigations) | 1 (2) | 4 (6)
Blood bilirubin increased (Investigations) | 1 (3) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (5) | 1 (1)
International Normalized Ratio (INR) increased (Investigations) | 2 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (10) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (6) | 8 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other (Endocrine disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT03136055/Prot_SAP_000.pdf